CLINICAL TRIAL: NCT02815150
Title: Safety and Effectiveness of Oral Administration of 5% Glucose Solution 250ml 2-3 Hours Before Surgery in Gastric Cancer Patients for Elective Radical Resection
Brief Title: Safety of 250ml Preoperative Carbohydrate Drink in Gastric Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: The First Affiliated Hospital of the Fourth Military Medical University (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Dongjie Yang, Associate professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016018
Record Dates: First submitted 2016-06-05; First posted 2016-06-28 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2019-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Treatment group (Experimental): Preoperative oral carbohydrate drink: patients drink 5% glucose solution 250ml 2-3 hours before surgery.
  Interventions: Dietary Supplement: preoperative oral carbohydrate drink
- Control group (No Intervention): Patients undergo 6-8 hours of preoperative fasting.

INTERVENTIONS:
Dietary Supplement: preoperative oral carbohydrate drink — 5% glucose solution 250ml 2-3 hours before surgery
  Arms: Treatment group

SUMMARY:
This study aims to assess the impact of preoperative oral carbohydrate drink on gastric emptying and PH of gastric fluid in gastric cancer patients directly. Furthermore, investigators aim to evaluate the safety and effectiveness of preoperative oral carbohydrate in elective gastric cancer surgery, providing direct evidence for clinical practice.

DETAILED DESCRIPTION:
In clinic, administration of oral carbohydrate 2-3 hours before surgery has been widely applied in elective colorectal surgery. However, no direct evidence has been showed that whether it is safe to do so in gastric cancer patients who are fit for elective radical gastric resection.

This study aims to discuss the impact and safety of oral administration of 5% glucose solution 250ml 2-3 hours before elective gastric cancer surgery. It is an equivalence study, which refers to a single-center, prospective, single blind, and randomized controlled study design. Eighty-eight patients with gastric adenocarcinoma are going to be enrolled in the study, who will be allocated into control or treatment group. Patients in control group follow the traditional routine of 6-8 hours preoperative fasting, while those in the treatment group will orally intake 250ml 5% glucose solution 2-3 hours before surgery. The primary end-point is the preoperative gastric residual volume. The secondary end-points include preoperative PH of gastric fluid, assessment of perioperative psychosomatic conditions, rate of perioperative complications, level of insulin sensitivity, recovery of bowel function, and the length of hospital stay, etc.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Histologically confirmed gastric adenocarcinoma
* Tumor of cT2-4aN0-2 in preoperative gastroscopy, endoscopic ultrasound, and/or abdominal computed tomography
* Fit for elective radical resection
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* American Society of Anesthesiology (ASA) status I to III
* Body mass index (BMI) of 17.5-27.5 kg/m2 .Patient agreed to participate this trial through informed consent.

Exclusion Criteria:

* Symptoms of pyloric obstruction
* Impaired bowel function, using drugs disturbing gastric secretion and gastric emptying
* History of gastric resection
* History of gastric cancer treatment
* History of major abdominal operation, or diffuse peritonitis
* Diabetes or impaired glucose tolerance, or with abnormality in other endocrine hormones
* Potential difficult airway as evaluated by anesthesiologist
* Pregnancy or breastfeeding were excluded in this trial .Patients would also be excluded if the following circumstances occurred: (1) failure of endotracheal intubation; (2) failure of intra-operative gastroscopy; or (3) irresectable tumor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-04-01; Primary Completion 2019-01-06 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
preoperative gastric residual volume of gastric fluid | 20-30 minutes before the surgery
  After anesthesia induction with 100-120mg propofol and 0.5 mg/kg rocuronium bromide and tracheal intubation, keep the patient in left lateral decubitus position. Insert the gastroscope ( Olympus 260) and perform complete suction of gastric fluid under direct vision with the suction apparatus connecting to the sterile airtight collector. Measure the volume of the gastric fluid in collector with a cylindrical measuring cup, accurate to 0.1ml. Repeat it and then take an average.

SECONDARY OUTCOMES:
Preoperative PH of gastric fluid | 20-30 minutes before the surgery
  bromide and tracheal intubation, keep the patient in left lateral decubitus position. Insert the gastroscope ( Olympus 260) and perform complete suction of gastric fluid under direct vision with the suction apparatus connecting to the sterile airtight collector. Inject 1ml clear gastric fluid into a vacuum drying tube by syringe and detect the PH value with the Delta 320 PH Detector twice and calculate the average value.
Preoperative thirsty/hungry scoring | 1 hour before the surgery
  Visual analogue scale with the score 0-10, 0 the least, 10 the most
Rate of perioperative complications | 7-8 days
  Including surgery-specific complications, such as bleeding, anastomosis leakage, and non-surgery-specific ones, such as lung infection, urinary tract infection, etc.
Recovery of bowel function | 3-7 days
  Record the time, by using postoperative days(POD), to first flatus, first stool and the time to endure semifluid diet
Perioperative insulin sensitivity | 8 days
  Quantitative Insulin Sensitivity Check Index, QUICKI = 1/ [ log ( I0) + log (G0) ]，I0 is the fasting insulin value, G0 is the fasting blood glucose value。
Length of hospital stay | 2-3 weeks
  Post operative hospital stay
Readmission rate within 30 days post operation | 1 month after surgery
  Readmission for any reason within 30 days after the surgery.
Reoperation rate within 30 days post operation | 1 month after surgery
  Reoperation that happens within 30 days after the primary surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dongjie Yang, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No